CLINICAL TRIAL: NCT01443026
Title: R01 CA90759: The Effects of Lycopene on High Risk Prostatic Tissue
Brief Title: The Effects of Lycopene on High Risk Prostatic Tissue
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Peter Gann, Professor and Director, Division of Pathology Research, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2005-0828; R01CA090759 (NIH)
Record Dates: First submitted 2011-09-27; First posted 2011-09-29 (Estimated); Results first posted 2015-06-04 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Intraepithelial Prostatic Neoplasia; Prostatic Neoplasms
Keywords: Intraepithelial Prostatic Neoplasia; Prostatic neoplasms; Male urogenital disease; Prostate
MeSH Terms: conditions — Prostatic Intraepithelial Neoplasia; Prostatic Neoplasms; Male Urogenital Diseases | interventions — Lycopene; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lycopene (Experimental): Lycopene 30 mg/day
  Interventions: Drug: Lycopene 30mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lycopene 30mg — Lycopene 30 mg.
  Other Names: Lyco-Mato
  Arms: Lycopene
Drug: Placebo — Placebo
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The purpose of this research study is to compare the effects of a lycopene supplement made from tomatoes to a placebo (a capsule with no active ingredients) in men who have abnormal cells in the prostate, but have not yet had cancer detected. This study will allow us to see if taking lycopene for six months leads to favorable changes in abnormal prostate tissue and in chemicals measured in the blood that go along with a higher risk of developing cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Have a history of prostate biopsy indicating HGPIN without cancer within 2 years prior to registration. At least 4 weeks must have elapsed between the last biopsy and the biopsy used for baseline data.
* Have an AUA symptom score <=25 at time of registration.
* Refrain from taking lycopene, selenium, vitamin E, or other antioxidant supplements within 1 month of randomization. Participants must agree to refrain from taking non-study dietary supplements while on study
* Refrain from taking exogenous hormones, drugs affecting hormone metabolism, or specified non-prescription substances (e.g. saw palmetto, PC-Spes) taken to affect the prostate within 1 month of registration. Patients must also agree to refrain from taking the non-prescription substances while on study
* Be willing to limit intake of lycopene-containing foods while on study
* Have no prior cancer (except basal cell or squamous cell skin cancer) or complete remission for at least 5 years
* Be ambulatory, capable of self-care and able to carry out light or sedentary work
* Have a dietary fat intake of 23-48% of calories
* Participant's physician recommends repeat biopsy 4-6 months after randomization

Exclusion Criteria:

* No repeat biopsy planned
* Not willing to change diet
* Have a diagnosis of prostate cancer

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2006-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter H Gann, MD, ScD, Principal Investigator — University of Illinois at Chicago
Locations (2):
- United States (2):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Jesse Brown VA Medical Center, Chicago, Illinois

REFERENCES:
- [Background] Clinton SK, Emenhiser C, Schwartz SJ, Bostwick DG, Williams AW, Moore BJ, Erdman JW Jr. cis-trans lycopene isomers, carotenoids, and retinol in the human prostate. Cancer Epidemiol Biomarkers Prev. 1996 Oct;5(10):823-33. PMID 8896894
- [Background] Pastori M, Pfander H, Boscoboinik D, Azzi A. Lycopene in association with alpha-tocopherol inhibits at physiological concentrations proliferation of prostate carcinoma cells. Biochem Biophys Res Commun. 1998 Sep 29;250(3):582-5. doi: 10.1006/bbrc.1998.9351. PMID 9784387
- [Background] Giovannucci E. Tomatoes, tomato-based products, lycopene, and cancer: review of the epidemiologic literature. J Natl Cancer Inst. 1999 Feb 17;91(4):317-31. doi: 10.1093/jnci/91.4.317. PMID 10050865
- [Background] Jain MG, Hislop GT, Howe GR, Ghadirian P. Plant foods, antioxidants, and prostate cancer risk: findings from case-control studies in Canada. Nutr Cancer. 1999;34(2):173-84. doi: 10.1207/S15327914NC3402_8. PMID 10578485
- [Background] Giovannucci E, Ascherio A, Rimm EB, Stampfer MJ, Colditz GA, Willett WC. Intake of carotenoids and retinol in relation to risk of prostate cancer. J Natl Cancer Inst. 1995 Dec 6;87(23):1767-76. doi: 10.1093/jnci/87.23.1767. PMID 7473833
- [Background] Bostwick DG, Shan A, Qian J, Darson M, Maihle NJ, Jenkins RB, Cheng L. Independent origin of multiple foci of prostatic intraepithelial neoplasia: comparison with matched foci of prostate carcinoma. Cancer. 1998 Nov 1;83(9):1995-2002. doi: 10.1002/(sici)1097-0142(19981101)83:93.0.co;2-2. PMID 9806659
- [Background] Kley HK. [Therapy of Cushing's syndrome. Critical evaluation of therapeutic measures]. Hippokrates. 1978 Feb;49(1):97-100. No abstract available. German. PMID 632120

RESULTS

PARTICIPANT FLOW:
Groups:
- Lycopene: Lycopene 30 mg/day until clinically-indicated repeat biopsy performed (approximately 6 months)
  Lycopene 30 mg or Placebo: Taken until clinically-indicated repeat biopsy performed (approximately 6 months)
- Placebo: Placebo taken until clinically-indicated repeat biopsy performed (approximately 6 months)
  Lycopene 30 mg or Placebo: Taken until clinically-indicated repeat biopsy performed (approximately 6 months)
Period: Overall Study
Arm/Group | Lycopene | Placebo
Started | 29 | 37
Completed | 26 | 32
Not Completed | 3 | 5
Not completed — Physician Decision | 1 | 0
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Lycopene: Lycopene 30 mg/day until clinically-indicated repeat biopsy performed (approximately 6 months)
- Placebo: Placebo taken until clinically-indicated repeat biopsy performed (approximately 6 months)
- Total: Total of all reporting groups
Arm/Group | Lycopene | Placebo | Total
Number analyzed (Participants) | 26 | 32 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (8.3) | 67.1 (8.1) | 65.2 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 26 | 32 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 9 | 15
  White | 19 | 23 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 32 | 58

OUTCOME MEASURES:

1. Primary Outcome: Tissue Biomarkers
Description: We will use conventional immunohistochemistry and computer-based image analysis to test the hypothesis that the lycopene supplements alter the expression of proteins marking the status of proliferation, differentiation, cell regulation and apoptosis in high-risk tissue.
Time Frame: baseline and 6 months
Reporting Status: Not Posted

2. Primary Outcome: Changes in Serum Biomarkers
Description: Change in serum lycopene, umol/L
Time Frame: baseline and 6 months
Measure: Mean (Full Range); unit: umol/L
Arm/Group | Lycopene | Placebo
Number analyzed (Participants) | 26 | 32
umol/L | .55 [-0.7 to 1.6] | -0.29 [-1.1 to 0.6]

3. Secondary Outcome: Changes in Nuclear Morphometry
Description: We will use a computerized image analysis system designed for the chemoprevention setting to test the hypothesis that the antioxidants cause a favorable change in a nuclear morphometry index based on nuclear size, shape and chromatin texture.
Time Frame: baseline and 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Lycopene | Placebo
Serious Adverse Events (participants affected / at risk) | 0/26 | 1/32
Other Adverse Events (participants affected / at risk) | 0/26 | 1/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lycopene (N=26) | Placebo (N=32)
death (Cardiac disorders) | 0 (0) | 1 (1) — Patient died four days after randomization from CAD. Patient was on placebo. Event was unrelated to study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lycopene (N=26) | Placebo (N=32)
increased urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No